CLINICAL TRIAL: NCT01078376
Title: A Comparative Single-Dose Pharmacokinetic and Safety Study of TAK-491 Between Infants, Children, and Adolescents With Hypertension and Healthy Adults
Brief Title: A Comparative Single-Dose Pharmacokinetic (PK) and Safety Study of Azilsartan Medoxomil in Children With Hypertension and in Healthy Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision (see below)
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: TAK-491_109; 2009-013165-25 (EudraCT Number); U1111-1113-4416 (Registry Identifier: WHO)
Record Dates: First submitted 2010-02-26; First posted 2010-03-02 (Estimated); Results first posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-06

CONDITIONS: Hypertension
Keywords: Pediatrics; Blood Pressure, High; Drug Therapy
MeSH Terms: conditions — Hypertension | interventions — azilsartan medoxomil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1: Healthy Adults (18 years to 45 years old) (Experimental): Azilsartan medoxomil 80 mg, tablets, orally, one day only
  Interventions: Drug: Azilsartan medoxomil (TAK-491)
- Cohort 1: Adolescents (≥12 to <17 years old) (Experimental): Azilsartan medoxomil 20 mg to 60 mg (based on participant weight), tablets, orally, one day only
  Interventions: Drug: Azilsartan medoxomil (TAK-491)
- Cohort 2: Children (≥6 to <12 years old) (Experimental): Azilsartan medoxomil 20 mg to 60 mg (based on participant weight), tablets, orally, one day only
  Interventions: Drug: Azilsartan medoxomil (TAK-491)
- Cohort 3: Children (≥1 to <6 years old) (Experimental): Azilsartan medoxomil 0.66 mg/kg participant body weight, granules, reconstituted orally, one day only
  Interventions: Drug: Azilsartan medoxomil (TAK-491)

INTERVENTIONS:
Drug: Azilsartan medoxomil (TAK-491) — Azilsartan medoxomil 80 mg, tablets, orally, one day only
  Other Names: TAK-491
  Arms: Cohort 1: Healthy Adults (18 years to 45 years old)
Drug: Azilsartan medoxomil (TAK-491) — Azilsartan medoxomil 20 mg to 60 mg (based on participant weight), tablets, orally, one day only
  Other Names: TAK-491
  Arms: Cohort 1: Adolescents (≥12 to <17 years old)
Drug: Azilsartan medoxomil (TAK-491) — Azilsartan medoxomil 20 mg to 60 mg (based on participant weight), tablets, orally, one day only
  Other Names: TAK-491
  Arms: Cohort 2: Children (≥6 to <12 years old)
Drug: Azilsartan medoxomil (TAK-491) — Azilsartan medoxomil 0.66 mg/kg participant body weight, granules, reconstituted orally, one day only
  Other Names: TAK-491
  Arms: Cohort 3: Children (≥1 to <6 years old)

SUMMARY:
The purpose of this study was to assess the pharmacokinetics (PK) and safety of a single dose of azilsartan medoxomil in children with hypertension, and comparative PK in healthy adults.

DETAILED DESCRIPTION:
Within the past 10 years, the incidence of high blood pressure (hypertension) in children and adolescents has increased all over the world. This increase is connected in part to a growing number of people who are overweight and do not eat right or exercise enough. In younger children though, high blood pressure is a common consequence of underlying diseases, such as renal diseases.

This study looked at a blood pressure medicine called TAK-491 (azilsartan medoxomil) to see how it works in children who have hypertension. Azilsartan medoxomil is a prodrug that converts into TAK-536 (azilsartan), a blood pressure lowering medicine that had not been tested in children.

To be eligible to take part in this study, children with a diagnosis of hypertension (primary or secondary) must have been between the ages of 1 year and 16 years old (up to their 17th birthday). Each child was given one dose of azilsartan medoxomil, followed by a number of blood tests and assessments within 24 hours after taking azilsartan medoxomil to see how the medication is working. Adults who do not have hypertension also took part in this study to provide comparison.

This study took place in 9 sites in the UK and USA. A total of 20 children with hypertension and 9 adults without hypertension participated in this study.

This study lasted about 43 days. This included a 28 day screening period, a 2 day treatment phase and a follow up period. Each participant taking part in this study may have been requested to remain in a hospital for one overnight stay during the course of the study. Each participant was contacted by telephone 6 days and 15 days after taking azilsartan medoxomil.

Takeda has decided to close Cohort 3 (participants between 1 and 6 years of age with hypertension) enrollment early and end this study with the agreement of both the US Food and Drug Administration (FDA) and the Pediatric Committee (PDCO) at the European Medicines Agency. Requests to the FDA and PDCO were submitted to close the study without completion of enrollment in Cohort 3 due to difficulty enrolling this particular patient population. Takeda proposed an alternative option to collect PK data in this age subset by utilizing PK modeling to determine the appropriate doses in children 1-5 years of age in lieu of completing Cohort 3. The FDA and PDCO agreed with this approach.

ELIGIBILITY:
Inclusion Criteria:

For Pediatric Participants:

Must have a diagnosis of hypertension (SBP and/or DBP ≥95th percentile for age/gender/height).

* For Cohorts 1 and 2 only, is within the weight range of 20 kg (44 pounds) to 100 kg (220 pounds), inclusive, at Screening.
* For Cohort 3 only, weighs at least 8.0 kg (17.6 pounds) at Screening.
* Participants greater than or equal to 6 years of age must have the ability to swallow a tablet of the size 6.0 millimeter diameter and 3.5 millimeter thickness.
* Has no known history of hepatitis B, hepatitis C, and human immunodeficiency virus.
* For Cohort 3 only, may be renal transplant patient if all other inclusion and none of the exclusion criteria are met, along with additional criteria.
* Must have been at a constant weight, or expected weight gain for that particular age, for 30 days with no change to the dose of their diuretic drugs.

For Healthy Adult Participants:

* Weighs at least 50 kilograms (110 pounds) and has a screening body mass index between 18 and 32 kilograms/m2, inclusive.
* Is in good health as determined by the physician
* Has a negative test result for hepatitis B surface antigen and antibody to hepatitis C virus, and has no known history of human immunodeficiency virus.
* Must have a negative urine test result for selected substances of abuse .
* Has a diastolic blood pressure between 60 and 90 mm Hg, inclusive, and a systolic blood pressure between 100 and 140 mm Hg, inclusive.

For All Participants:

* Females of child bearing potential who are sexually active, as well as sexually active male participants, agree to routinely use adequate contraception from Screening until 30 days after receiving the last dose of study medication.
* Has clinical laboratory results within the reference range for the testing laboratory unless the results are deemed not clinically significant by the investigator.

Exclusion Criteria:

For Pediatric Participants:

* Is currently treated with more than 2 antihypertensive agents.
* Has sitting trough clinic systolic blood pressure greater than 15 mm Hg or diastolic blood pressure greater than 10 mm Hg above the 99th percentile for age, gender, and height at Check-in .
* Has renovascular disease affecting both kidneys or a solitary kidney, dialysis treatment, severe nephrotic syndrome and not in remission.
* For Cohort 1 and 2 only, a previous renal transplant.
* Has a creatinine clearance less than 30 mL/min/1.73 m2.

For all participants:

* Has previously received azilsartan or azilsartan medoxomil.
* Has a known hypersensitivity or allergy to any angiotensin type II receptor blockers or to any of the excipients in the azilsartan medoxomil formulation to be taken.
* Has a history or clinical manifestations of severe cardiovascular disease, psychiatric disease, and any conditions that would interfere with gastrointestinal absorption.
* Has hemodynamically significant left ventricular outflow obstruction due to aortic valvular disease, cardiomyopathy, or uncorrected coarctation of the aorta.
* Has been diagnosed with malignant or accelerated hypertension.
* Has severe hepatic impairment.
* Has a serum albumin less than 2.5 g/dL.
* Has a glycosylated hemoglobin value greater than 8.5%.
* Has alanine aminotransferase, aspartate aminotransferase greater than 2 times the upper limit of normal, or total bilirubin greater than 1.5 times the upper limit of normal, active liver disease, or jaundice.
* Has hyperkalemia as defined by the laboratory normal reference range or any pertinent electrolyte disorders.
* Is participating in another investigational study or has taken an investigational drug within 30 days prior to Check-in .
* Has a history of drug abuse or a history of alcohol abuse within 1 year prior to study Check-in.
* Has a history of abdominal surgery or thoracic or nonperipheral vascular surgery within 6 months prior to study Check-in.
* Has a history of cancer, other than basal cell carcinoma or stage I squamous cell carcinoma of the skin that has not been in remission for at least 5 years prior to study Check-in.
* Has taken any cytotoxic drugs within 12 months prior to study Check-in .
* Has a history or presence of a clinically significant abnormal 12-lead electrocardiogram as determined by the investigator or sponsor/designee.
* Has poor peripheral venous access.
* Has any other condition or prior therapy that, in the opinion of the investigator, would make the participant unsuitable for the study.
* Has taken or requires the use of any medications, supplements, or food products within the stated time periods, including:

  * Pediatric participants taking angiotensin-converting enzyme inhibitors and other angiotensin II receptor blockers will be required to withhold these medications from the morning of Day -1 until the 24 hour pharmacokinetic sample is completed on Day 2.
  * Only pediatric participants will be allowed to take medications for primary renal or urologic conditions or hypertension as long as they have been on a stable dose of their medication for at least 30 days prior to Check-in (Day -1) and those medications are not potent cytochrome P-450 inhibitors or inducers.
  * Nutraceuticals including herbal or dietary preparations such as ginseng, kava kava, and ginkgo biloba.
  * Over-the-counter medications.
  * Vitamin supplements except for pediatric participants only.
  * Alcohol-containing products.
  * Products that contain caffeine or xanthine-related compounds.
  * Foods or beverages containing grapefruit juice or Seville-type oranges.

Ages: 1 Year to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2010-05; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (8):
- United States (4):
  - Little Rock, Arkansas
  - Atlanta, Georgia
  - Louisville, Kentucky
  - Toledo, Ohio
- United Kingdom (4):
  - Birmingham, England
  - Bristol, England
  - London, England
  - Manchester, England

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 6 sites in the United States and 3 sites in the United Kingdom from 10 May 2010 to 10 July 2013.
Pre-assignment Details: Children between the ages of 1 to 16 years (including up to their 17th birthday) with hypertension and gender-matched healthy adults aged 18 to 45 years, inclusive, were enrolled in 1 of 3 cohorts.
Groups:
- Cohort 1: Healthy Adults: Azilsartan medoxomil 80 mg, tablets, orally, one day only
- Cohort 1: Adolescents (≥12 to <17 Years Old) 40-60 mg: Azilsartan medoxomil 40-60 mg, tablets, orally, one day only. Dose regimen was based on body weight. Participants 40 to < 80 kg received a 40 mg dose and participants 80 to 100 kg received a 60 mg dose.
- Cohort 2: Children (≥6 to <12 Years Old) 20-60 mg: Azilsartan medoxomil 20-60 mg, tablets, orally, one day only. Dose regimen was based on body weight. Participants 20 to < 40 kg received a 20 mg dose, participants 40 to < 80 kg received a 40 mg dose and participants 80 to 100 kg received a 60 mg dose.
Period: Overall Study
Arm/Group | Cohort 1: Healthy Adults | Cohort 1: Adolescents (≥12 to <17 Years Old) 40-60 mg | Cohort 2: Children (≥6 to <12 Years Old) 20-60 mg | Cohort 3: Children (≥1 to <6 Years Old)
Started | 9 | 9 | 8 | 3
Completed | 9 | 9 | 8 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Healthy Adults | Cohort 1: Adolescents (≥12 to <17 Years Old) 40-60 mg | Cohort 2: Children (≥6 to <12 Years Old) 20-60 mg | Cohort 3: Children (≥1 to <6 Years Old) | Total
Number analyzed (Participants) | 9 | 9 | 8 | 3 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (7.78) | 14.2 (1.64) | 9.1 (2.10) | 4.7 (0.58) | 16.2 (9.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 5 | 2 | 11
  Male | 7 | 7 | 3 | 1 | 18
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 4 | 0 | 1 | 0 | 5
  Not Hispanic or Latino | 5 | 7 | 5 | 3 | 20
  Not Reported | 0 | 2 | 2 | 0 | 4
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 0 | 1 | 0 | 1
  Black or African American | 1 | 2 | 2 | 2 | 7
  White | 8 | 7 | 5 | 1 | 21
Height [Mean (Standard Deviation); unit: cm] | 172.6 (9.70) | 163.1 (11.72) | 138.6 (12.74) | 107.7 (11.06) | 153.6 (23.45)
Weight [Mean (Standard Deviation); unit: kg] | 74.64 (11.207) | 71.71 (15.512) | 48.50 (22.523) | 18.30 (4.026) | 60.69 (23.859)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.06 (3.345) | 27.22 (6.611) | 24.29 (8.327) | 15.67 (0.551) | 24.54 (6.625)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Time of Last Quantifiable Concentration (AUC[0-tlqc]) for TAK-536
Description: AUC(0-tlqc) is a measure of total plasma exposure to the drug from Time 0 to Time of the Last Quantifiable Concentration (AUC[0-tlqc]).
Time Frame: Day 1
Population: Pharmacokinetic Set; Results are presented by individual dose for Cohorts 1 and 2.
Measure: Mean (Standard Deviation); unit: ng.hr/mL
Groups:
- Cohort 1: Adolescents (≥12 to <17 Years Old) 60 mg; Cohort 2: Children (≥6 to <12 Years Old) 60 mg: Azilsartan medoxomil 60 mg, tablets, orally, one day only
- Cohort 1: Adolescents (≥12 to <17 Years Old) 40 mg; Cohort 2: Children (≥6 to <12 Years Old) 40 mg: Azilsartan medoxomil 40 mg, tablets, orally, one day only
- Cohort 2: Children (≥6 to <12 Years Old) 20 mg: Azilsartan medoxomil 20 mg, tablets, orally, one day only
Arm/Group | Cohort 1: Healthy Adults | Cohort 1: Adolescents (≥12 to <17 Years Old) 60 mg | Cohort 1: Adolescents (≥12 to <17 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 60 mg | Cohort 2: Children (≥6 to <12 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 20 mg | Cohort 3: Children (≥1 to <6 Years Old)
Number analyzed (Participants) | 9 | 2 | 6 | 1 | 4 | 3 | 3
ng.hr/mL | 40613 (9609.6) | 23889 (5383.8) | 17423 (3559.7) | 16056 (NA) — Standard deviation can not be calculated for 1 participant. | 22556 (5792.6) | 18691 (5489.9) | 16963 (4948.4)

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Time of Last Quantifiable Concentration (AUC[0-tlqc]) for TAK-536 Metabolite M-II.
Description: as for outcome 1
Time Frame: Day 1
Population: Pharmacokinetic Set; Results are presented by individual dose for Cohorts 1 and 2.
Measure: Mean (Standard Deviation); unit: ng.hr/mL
Arm/Group | Cohort 1: Healthy Adults | Cohort 1: Adolescents (≥12 to <17 Years Old) 60 mg | Cohort 1: Adolescents (≥12 to <17 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 60 mg | Cohort 2: Children (≥6 to <12 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 20 mg | Cohort 3: Children (≥1 to <6 Years Old)
Number analyzed (Participants) | 9 | 2 | 6 | 1 | 4 | 3 | 3
ng.hr/mL | 11563 (3106.5) | 7409 (78.6) | 7428 (2120.7) | 7392 (NA) — Standard deviation can not be calculated for 1 participant. | 7929 (3502.6) | 9130 (1338.3) | 7285 (3626.0)

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC[0-inf]) for TAK-536
Description: Area under the plasma concentration-time curve from time 0 to infinity, calculated as AUC(0-inf)=AUC(0-tlqc) + Clast/λz.
Time Frame: Day 1
Population: Pharmacokinetic Set; Results are presented by individual dose for Cohorts 1 and 2.
Measure: Mean (Standard Deviation); unit: ng.hr/mL
Arm/Group | Cohort 1: Healthy Adults | Cohort 1: Adolescents (≥12 to <17 Years Old) 60 mg | Cohort 1: Adolescents (≥12 to <17 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 60 mg | Cohort 2: Children (≥6 to <12 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 20 mg | Cohort 3: Children (≥1 to <6 Years Old)
Number analyzed (Participants) | 9 | 2 | 6 | 1 | 4 | 3 | 3
ng.hr/mL | 44820 (11680.7) | 26411 (6703.1) | 18686 (3720.4) | 16563 (NA) — Standard deviation can not be calculated for 1 participant. | 23792 (6157.0) | 19543 (6181.1) | 17771 (5263.1)

4. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC[0-inf]) for TAK-536 Metabolite M-II
Description: Area under the plasma concentration-time curve from time 0 to infinity, calculated as AUC(0-inf)=AUC(0-tlqc) + Clast/λz.
Time Frame: Day 1
Population: Pharmacokinetic Set; Results are presented by individual dose for Cohorts 1 and 2.
Measure: Mean (Standard Deviation); unit: ng.hr/mL
Arm/Group | Cohort 1: Healthy Adults | Cohort 1: Adolescents (≥12 to <17 Years Old) 60 mg | Cohort 1: Adolescents (≥12 to <17 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 60 mg | Cohort 2: Children (≥6 to <12 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 20 mg | Cohort 3: Children (≥1 to <6 Years Old)
Number analyzed (Participants) | 9 | 2 | 6 | 1 | 4 | 3 | 3
ng.hr/mL | 19188 (6766.0) | 10596 (1168.8) | 12532 (3905.3) | 8961 (NA) — Standard deviation can not be calculated for 1 participant. | 11387 (5440.7) | 14230 (3419.6) | 9477 (4659.6)

5. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for TAK-536
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Day 1
Population: Pharmacokinetic Set; Results are presented by individual dose for Cohorts 1 and 2.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: Healthy Adults | Cohort 1: Adolescents (≥12 to <17 Years Old) 60 mg | Cohort 1: Adolescents (≥12 to <17 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 60 mg | Cohort 2: Children (≥6 to <12 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 20 mg | Cohort 3: Children (≥1 to <6 Years Old)
Number analyzed (Participants) | 9 | 2 | 6 | 1 | 4 | 3 | 3
ng/mL | 5699 (1346.1) | 3245 (106.1) | 2512 (701.6) | 2810 (NA) — Standard deviation can not be calculated for 1 participant. | 3858 (1363.0) | 2960 (364.3) | 3320 (656.0)

6. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for TAK-536 Metabolite M-II
Description: as for outcome 5
Time Frame: Day 1
Population: Pharmacokinetic Set; Results are presented by individual dose for Cohorts 1 and 2.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: Healthy Adults | Cohort 1: Adolescents (≥12 to <17 Years Old) 60 mg | Cohort 1: Adolescents (≥12 to <17 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 60 mg | Cohort 2: Children (≥6 to <12 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 20 mg | Cohort 3: Children (≥1 to <6 Years Old)
Number analyzed (Participants) | 9 | 2 | 6 | 1 | 4 | 3 | 3
ng/mL | 736 (241.6) | 480 (74.2) | 535 (200.2) | 514 (NA) — Standard deviation can not be calculated for 1 participant. | 561 (211.7) | 561 (40.3) | 488 (212.2)

7. Primary Outcome: Time to Reach Cmax (Tmax) for TAK-536
Description: Tmax: Time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax, as observed on Day 1.
Time Frame: Day 1
Population: Pharmacokinetic Set; Results are presented by individual dose for Cohorts 1 and 2.
Measure: Median (Full Range); unit: hr
Arm/Group | Cohort 1: Healthy Adults | Cohort 1: Adolescents (≥12 to <17 Years Old) 60 mg | Cohort 1: Adolescents (≥12 to <17 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 60 mg | Cohort 2: Children (≥6 to <12 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 20 mg | Cohort 3: Children (≥1 to <6 Years Old)
Number analyzed (Participants) | 9 | 2 | 6 | 1 | 4 | 3 | 3
hr | 2.00 (0.8819) [2.00 to 4.00] | 2.01 (0.0118) [2.00 to 2.02] | 2.00 (0.4082) [1.00 to 2.00] | 2.00 (NA) [NA to NA] — Standard deviation or range cannot be calculated for 1 participant. | 2.00 (2.2043) [1.05 to 6.00] | 2.00 (0.0096) [1.98 to 2.00] | 1.00 (0.0000) [1.00 to 1.00]

8. Primary Outcome: Time to Reach Cmax (Tmax) for TAK-536 Metabolite M-II
Description: Tmax: Time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax, as observed on Day 1.
Time Frame: Day 1
Population: Pharmacokinetic Set; Results are presented by individual dose for Cohorts 1 and 2.
Measure: Median (Full Range); unit: hr
Arm/Group | Cohort 1: Healthy Adults | Cohort 1: Adolescents (≥12 to <17 Years Old) 60 mg | Cohort 1: Adolescents (≥12 to <17 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 60 mg | Cohort 2: Children (≥6 to <12 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 20 mg | Cohort 3: Children (≥1 to <6 Years Old)
Number analyzed (Participants) | 9 | 2 | 6 | 1 | 4 | 3 | 3
hr | 6.00 (1.4227) [4.00 to 8.00] | 5.00 (1.4142) [4.00 to 6.00] | 6.00 (0.8256) [4.00 to 6.10] | 6.00 (NA) [NA to NA] — Standard deviation or range cannot be calculated for 1 participant. | 4.03 (1.9890) [4.00 to 8.00] | 4.00 (2.3094) [4.00 to 8.00] | 6.0 (0.0000) [6.00 to 6.00]

9. Primary Outcome: Terminal Elimination Half-life (T1/2) for TAK-536
Description: Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Time Frame: Day 1
Population: Pharmacokinetic Set; Results are presented by individual dose for Cohorts 1 and 2.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Cohort 1: Healthy Adults | Cohort 1: Adolescents (≥12 to <17 Years Old) 60 mg | Cohort 1: Adolescents (≥12 to <17 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 60 mg | Cohort 2: Children (≥6 to <12 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 20 mg | Cohort 3: Children (≥1 to <6 Years Old)
Number analyzed (Participants) | 9 | 2 | 6 | 1 | 4 | 3 | 3
hr | 7.35 (1.083) | 7.74 (0.621) | 5.76 (1.158) | 5.07 (NA) — Standard deviation can not be calculated for 1 participant. | 5.75 (0.760) | 5.37 (0.922) | 4.59 (1.627)

10. Primary Outcome: Terminal Elimination Half-life (T1/2) for TAK-536 Metabolite M-II
Description: Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Time Frame: Day 1
Population: Pharmacokinetic Set; Results are presented by individual dose for Cohorts 1 and 2.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Cohort 1: Healthy Adults | Cohort 1: Adolescents (≥12 to <17 Years Old) 60 mg | Cohort 1: Adolescents (≥12 to <17 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 60 mg | Cohort 2: Children (≥6 to <12 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 20 mg | Cohort 3: Children (≥1 to <6 Years Old)
Number analyzed (Participants) | 9 | 2 | 6 | 1 | 4 | 3 | 3
hr | 16.60 (6.870) | 12.78 (2.915) | 14.00 (2.414) | 8.50 (NA) — Standard deviation can not be calculated for 1 participant. | 11.56 (3.314) | 13.97 (2.983) | 10.35 (2.770)

11. Primary Outcome: Apparent Oral Clearance (CL/F) for TAK-536
Description: CL/F is apparent clearance of the drug from the plasma, expressed in L/hr.
Time Frame: Day 1
Population: Pharmacokinetic Set; Results are presented by individual dose for Cohorts 1 and 2.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Cohort 1: Healthy Adults | Cohort 1: Adolescents (≥12 to <17 Years Old) 60 mg | Cohort 1: Adolescents (≥12 to <17 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 60 mg | Cohort 2: Children (≥6 to <12 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 20 mg | Cohort 3: Children (≥1 to <6 Years Old)
Number analyzed (Participants) | 9 | 2 | 6 | 1 | 4 | 3 | 3
L/hr | 1.52 (0.414) | 1.88 (0.477) | 1.78 (0.411) | 2.90 (NA) — Standard deviation can not be calculated for 1 participant. | 1.43 (0.427) | 0.87 (0.232) | 0.54 (0.134)

12. Primary Outcome: Total Amount of Drug Excreted in Urine From Time 0 to 24 Hours Postdose (Ae[0-t]) (for Cohorts 1 and 2 Urine Pharmacokinetic Endpoint for TAK-536)
Time Frame: Day 1
Population: Pharmacokinetic Set; Results are presented by individual dose for Cohorts 1 and 2.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Cohort 1: Healthy Adults | Cohort 1: Adolescents (≥12 to <17 Years Old) 60 mg | Cohort 1: Adolescents (≥12 to <17 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 60 mg | Cohort 2: Children (≥6 to <12 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 20 mg
Number analyzed (Participants) | 9 | 3 | 6 | 1 | 4 | 3
mg | 10.65 (4.673) | 4.56 (1.029) | 2.89 (0.936) | 4.59 (NA) — Standard deviation can not be calculated for 1 participant. | 3.63 (2.125) | 1.27 (0.580)

13. Primary Outcome: Total Amount of Drug Excreted in Urine From Time 0 to 24 Hours Postdose (Ae[0-t]) (for Cohorts 1 and 2 Urine Pharmacokinetic Endpoint for TAK-536 Metabolite M-II)
Time Frame: Day 1
Population: Pharmacokinetic Set; Results are presented by individual dose for Cohorts 1 and 2.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Cohort 1: Healthy Adults | Cohort 1: Adolescents (≥12 to <17 Years Old) 60 mg | Cohort 1: Adolescents (≥12 to <17 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 60 mg | Cohort 2: Children (≥6 to <12 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 20 mg
Number analyzed (Participants) | 9 | 3 | 6 | 1 | 4 | 3
mg | 6.60 (5.149) | 2.93 (0.582) | 2.73 (1.528) | 4.43 (NA) — Standard deviation can not be calculated for 1 participant. | 2.77 (1.197) | 1.48 (0.284)

14. Primary Outcome: Fraction of Unchanged Drug Excreted in Urine From 0 to 24 Hours Postdose (Fe%) (for Cohorts 1 and 2 Urine Pharmacokinetic Endpoint for TAK-536)
Description: Fe=[Ae(0-24)/dose]×100 (molecular weight adjusted for metabolites.
Time Frame: Day 1
Population: Pharmacokinetic Set; Results are presented by individual dose for Cohorts 1 and 2.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Cohort 1: Healthy Adults | Cohort 1: Adolescents (≥12 to <17 Years Old) 60 mg | Cohort 1: Adolescents (≥12 to <17 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 60 mg | Cohort 2: Children (≥6 to <12 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 20 mg
Number analyzed (Participants) | 9 | 3 | 6 | 1 | 4 | 3
percent | 16.65 (7.302) | 9.50 (2.144) | 9.04 (2.925) | 9.57 (NA) — Standard deviation can not be calculated for 1 participant. | 11.36 (6.639) | 7.94 (3.622)

15. Primary Outcome: Fraction of Unchanged Drug Excreted in Urine From 0 to 24 Hours Postdose (Fe%) (for Cohorts 1 and 2 Urine Pharmacokinetic Endpoint for TAK-536 Metabolite M-II)
Description: Fe=[Ae(0-24)/dose]×100 (molecular weight adjusted for metabolites.
Time Frame: Day 1
Population: Pharmacokinetic Set; Results are presented by individual dose for Cohorts 1 and 2.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Cohort 1: Healthy Adults | Cohort 1: Adolescents (≥12 to <17 Years Old) 60 mg | Cohort 1: Adolescents (≥12 to <17 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 60 mg | Cohort 2: Children (≥6 to <12 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 20 mg
Number analyzed (Participants) | 9 | 3 | 6 | 1 | 4 | 3
percent | 11.01 (8.581) | 6.55 (1.293) | 9.11 (5.094) | 9.85 (NA) — Standard deviation can not be calculated for 1 participant. | 9.22 (3.991) | 9.89 (1.896)

16. Primary Outcome: Renal Clearance (CLr) From 0 to 24 Hours Postdose (for Cohorts 1 and 2 Urine Pharmacokinetic Endpoint for TAK-536)
Description: Renal clearance, calculated as CLr=Ae(0-24)/AUC(0-24).
Time Frame: Day 1
Population: Pharmacokinetic Set; Results are presented by individual dose for Cohorts 1 and 2.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Cohort 1: Healthy Adults | Cohort 1: Adolescents (≥12 to <17 Years Old) 60 mg | Cohort 1: Adolescents (≥12 to <17 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 60 mg | Cohort 2: Children (≥6 to <12 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 20 mg
Number analyzed (Participants) | 9 | 2 | 6 | 1 | 4 | 3
L/hr | 0.28 (0.130) | 0.22 (0.051) | 0.17 (0.077) | 0.29 (NA) — Standard deviation can not be calculated for 1 participant. | 0.15 (0.069) | 0.07 (0.011)

17. Primary Outcome: Renal Clearance (CLr) From 0 to 24 Hours Postdose (for Cohorts 1 and 2 Urine Pharmacokinetic Endpoint for TAK-536 Metabolite M-II)
Description: Renal clearance, calculated as CLr=Ae(0-24)/AUC(0-24).
Time Frame: Day 1
Population: Pharmacokinetic Set; Results are presented by individual dose for Cohorts 1 and 2.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Cohort 1: Healthy Adults | Cohort 1: Adolescents (≥12 to <17 Years Old) 60 mg | Cohort 1: Adolescents (≥12 to <17 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 60 mg | Cohort 2: Children (≥6 to <12 Years Old) 40 mg | Cohort 2: Children (≥6 to <12 Years Old) 20 mg
Number analyzed (Participants) | 9 | 2 | 6 | 1 | 4 | 3
L/hr | 0.55 (0.309) | 0.37 (0.084) | 0.34 (0.146) | 0.60 (NA) — Standard deviation can not be calculated for 1 participant. | 0.36 (0.099) | 0.16 (0.022)

ADVERSE EVENTS:
Time Frame: A treatment-emergent adverse event (TEAE) had an onset occurring after the first dose of study medication and within 14 days after the last dose of study medication or, if an SAE, within 30 days after last dose of study medication.
Description: At each visit the investigator assessed whether any subjective adverse events have occurred and had to document any occurrence of adverse events and clinically significant abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cohort 1: Healthy Adults | Cohort 1: Adolescents (≥12 to <17 Years Old) 40-60 mg | Cohort 2: Children (≥6 to <12 Years Old) 20-60 mg | Cohort 3: Children (≥1 to <6 Years Old)
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/8 | 0/3
Other Adverse Events (participants affected / at risk) | 2/9 | 5/9 | 3/8 | 0/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Healthy Adults (N=9) | Cohort 1: Adolescents (≥12 to <17 Years Old) 40-60 mg (N=9) | Cohort 2: Children (≥6 to <12 Years Old) 20-60 mg (N=8) | Cohort 3: Children (≥1 to <6 Years Old) (N=3)
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Infusion site pain (General disorders) | 0 | 0 | 1 | 0
Infected bites (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was discontinued without complete enrollment of Cohort 3. Therefore, PK modeling will be used to determine the appropriate doses in children 1 to <6 years of age, in lieu of completing Cohort 3.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be made without Sponsor's prior written approval. Any proposed publication or presentation will be submitted to Sponsor for review 60 days in advance of publication. Institution will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for an additional 60 days to preserve intellectual property.